CLINICAL TRIAL: NCT02686671
Title: A New Diagnostic Clinical Test To Determine Responders To Subacromial Injection In Patients With Shoulder Impingement: A Case Series
Brief Title: The Pull Test To Determine Responders To Subacromial Injection In Patients With Shoulder Impingement
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L16-047
Record Dates: First submitted 2016-01-20; First posted 2016-02-19 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Bursitis; Injections; Shoulder Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Shoulder clinical examination testing — Shoulder clinical examination including resistive shoulder abduction with and without a humeral traction (Pull Test). Functional status will be measured using the Shoulder Pain and Disability Index (SPADI).

SUMMARY:
Shoulder pain is very common. People receive injections in their shoulder for their painful shoulder. However, investigators do not know which patient with shoulder pain responds best to an injection in the shoulder.

Investigators plan to use a "Pull Test" where the researcher will pull on the arm and resist shoulder movement to investigate if it helps to determine which patients have better pain relief with the shoulder injection.

The study will take place in Anchorage, Alaska. There will be two phases in the study. For each phase, the subjects will complete some questionnaires. Phase I "Reliability Testing" will test how consistent two licensed physical therapists are giving shoulder examination tests and the Pull Test. Phase II "Pull Test" will comprise shoulder examination findings, including the Pull Test, done before and after one shoulder injection performed as normal standard of care by a licensed physician.

For Phase I of the study, up to 20 patients treated for shoulder pain will be recruited from Advanced Physical Therapy. For Phase II of the study, up to 100 patients with shoulder pain scheduled to have a shoulder injection will be asked by an investigator if they wish to participate in the study until a number of 30 subjects qualify for the study. Phase II of the study will include shoulder tests before and about 20 minutes after the injection and a 4- to 7-day, as well as a 6-week, phone follow-up.

Statistics will be used to analyze the data.

DETAILED DESCRIPTION:
Background: Subacromial impingement syndrome (SAIS) is one of the most common causes of shoulder pain. The subacromial-subdeltoid (SAD) bursa is regarded as a common potential shoulder pain generator. Differentiating the specific acromio-humeral interval (AHI) tissues responsible for pain generation is challenging and no specific clinical examination testing exists to differentiate SAD bursa from the rotator cuff tendons as pain generators. Corticosteroid injection (CSI) within the AHI is a mainstay of treatment for SAD bursitis and rotator cuff tendinopathy. No study to date has examined a specific test associated with successful responsiveness from a CSI targeting the SAD bursa in the AHI in subjects with shoulder pain.

Purpose: To investigate (1) Phase I: the reliability of the shoulder examination tests and of the Pull Test; and (2) Phase II: if a positive shoulder traction test during resistive shoulder abduction, the "Pull Test", correlates with a successful outcome of an AHI CSI targeting the SAD bursa.

Aims: To evaluate: (1) the reliability of the Pull Test; (2) if a positive Pull Test correlates with successful pain and satisfaction outcomes immediately following, 4 to 7 days following, and 6 weeks following an AHI CSI targeting the SAD bursa in subjects with musculoskeletal shoulder pain (3) if a positive Pull Test correlates with a successful functional outcome 6 weeks following an AHI CSI targeting the SAD bursa in subjects with musculoskeletal shoulder pain and (4) the sensitivity, specificity, accuracy, positive and negative predictive values of the Pull Test to identify subjects with shoulder pain likely to successfully respond to an AHI CSI targeting the SAD bursa

Design: Methodological and exploratory correlational study.

Methods: Phase I (reliability testing): A sample of convenience of up to 20 subjects treated at Advanced Physical Therapy of Alaska for shoulder pain will be recruited to participate. Two licensed physical therapists will test the reliability of the shoulder examination tests and of the Pull Test. Phase II (Pull Test): A consecutive sample of convenience of subjects treated by physicians from Advanced Pain Centers of Alaska for musculoskeletal shoulder pain and scheduled for a subacromial CSI as part of their care will be asked to participate in the study. The study will end when a minimum of 30 subjects qualify for the research study. Those subjects agreeing to participate will then be evaluated using shoulder clinical examination including resistive shoulder abduction with and without a humeral traction (Pull Test). Functional status will be measured using the Shoulder Pain and Disability Index (SPADI). Following the CSI, one investigator blinded to the results of the pre-injection clinical examination will administer the clinical examination tests performed prior to the AHI CSI and record shoulder pain (NPRS) and subject satisfaction about the change in pain following the CSI. Subjects will then receive standardized home instructions. A 4- to 7-day follow-up phone call to determine shoulder pain (NPRS) and satisfaction and 6-week follow-up phone call to determine satisfaction and subjects' compliance to the home instructions, shoulder pain (NPRS) at rest and during arm elevation, SPADI score and subject satisfaction will be initiated.

Statistical Analysis: Reliability testing will be assessed using kappa and intraclass correlation coefficients. Validity testing of the Pull Test will be performed to determine the sensitivity, specificity, accuracy, negative and positive predictive values for the comparison of Pull Test outcome and the pain and functional changes observed following administration of the AHI CSI. Chi-square (2x2 contingency tables) and odds ratios will then be calculated to evaluate if the outcomes of the Pull Test (binary: positive versus negative) are correlated with successful pain and functional outcome changes following the AHI CSI (successful outcome, Yes versus No) immediately following, at 4- to 7-days following, and at 6-weeks following the AHI CSI.

ELIGIBILITY:
Inclusion Criteria: Subjects will be eligible for both phases of the study if they meet the following criteria:

* age 18 to 80 years
* demonstrate shoulder pain within the C5 distribution during resisted abduction between 2 and 10/10 on NRPS (Wainner et al 2003)
* demonstrate one or more positive tests out of the following clinical examination impingement tests: Neer's sign, Hawkins-Kennedy test, painful arc of arm elevation (Kessel & Watson 1977; Kelly et al 2010)
* painful resisted abduction of the shoulder (Kelly et al 2010)

Exclusion Criteria: Subjects will be excluded from the study for the following reasons:

* a large three-dimensional limitation of arm motion with any passive motion of the shoulder as compared to the contralateral side, to rule out adhesive capsulitis (Rundquist & Ludewig 2004; Tveita et al 2008)
* shoulder surgery within the last six months
* a CSI to the involved shoulder within the past three months
* presence of a systemic inflammatory condition
* presence of radiculopathy during active range of motion of the cervical spine (Wainner et al 2003)
* cervical spine as a current primary complaint over the shoulder
* pain reproduction during the Spurling Test (Henry et al 2002; Wainner et al 2003)
* inability to undergo a follow-up phone call
* neurological disorders such as multiple sclerosis, spinal cord injury or spinal cord tumors that would prevent subjects to elevate the arm above the head or perform shoulder movements against resistance
* pregnancy by self-report from the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive sample of convenience of subjects treated by physicians from Advanced Pain Centers of Alaska for musculoskeletal shoulder pain and scheduled for a subacromial CSI as part of their care will be asked to participate in the study. The study will end when a minimum of 30 subjects qualify for the research study.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Pain (NPRS) | 10-30 minutes
  Pain recording pre-injection
SPADI | Immediately pre-injection
  Shoulder function pre-injection
Pain (NPRS) | Immediately post-injection
  Pain recording immediately post-injection
Patient Satisfaction | Immediately post-injection
  Patient satisfaction immediately post-injection based on 5-point Likert Scale
Pain (NPRS) | 4-7 days
  Pain recording 4-7 days post-injection
Patient Satisfaction | 4-7 days
  Patient satisfaction 4-7 days post-injection based on 5-point Likert Scale
Pain (NPRS) | 6-weeks
  Pain recording 6-weeks post-injection
SPADI | 6-weeks
  Shoulder function 6-weeks post-injection
Patient Satisfaction | 6-weeks
  Patient satisfaction 6-weeks post-injection based on 5-point Likert Scale
Subjective Outcome of Success of Injection Assessed by Survey Question | Immediately post-injection
  Subjective assessment of successful outcome of shoulder injection using "Yes", "Unsure" and "No" as items
Subjective Outcome of Success of Injection Assessed by Survey Question | 4-7 days
  Subjective assessment of successful outcome of shoulder injection using "Yes", "Unsure" and "No" as items
Subjective Outcome of Success of Injection Assessed by Survey Question | 6-weeks
  Subjective assessment of successful outcome of shoulder injection using "Yes", "Unsure" and "No" as items

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Brismee, ScD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Advanced Physical Therapy, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02686671/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02686671/SAP_001.pdf